CLINICAL TRIAL: NCT05728151
Title: Comparing General Anesthesia With Single Injection Peribulbar Block With Articaine 4% vs Lidocaine 2% vs Mepivacaine 3 % for Prevention of Oculocardiac Reflex in Children Undergoing Strabismus Surgery : A Randomized Control Study
Brief Title: Comparing General Anesthesia With Single Injection Peribulbar Block With 3 Different Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIO2022
Record Dates: First submitted 2023-01-18; First posted 2023-02-14 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2022-02

CONDITIONS: Pediatric Squint Surgeries
MeSH Terms: interventions — Carticaine; Levobupivacaine; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- For group A (Experimental): Group A will be inducted as before in addition of giving a peribulbar block up to 5 ml ( according to the volume of the eye ) of Articaine 4 % with adrenaline 1/100000 mixed with 10IU of Hyaluronidase by a single injection technique: a 26/27 gauge needle will be inserted as far laterally as possible in the inferotemporal quadrant. Once the needle is under the globe, it will be directed along the orbital floor, passing the globe equator to a depth controlled by observing the needle/hub junction reaching the plane of the iris. After negative aspiration for blood, with the globe in primary gaze, and start injection and the injected volume will be guided by digital intraocular pressure.
  Interventions: Drug: Articaine and Epinephrine Only Product
- Group L (Experimental): General Anesthesia will be inducted as before in addition of giving a peribulbar block up to 5 ml ( according to the volume of the eye ) of Lidocaine 2%mixed with 10IU of Hyaluronidase by a single injection technique.
  Interventions: Drug: levobupivacaine
- Group M (Experimental): General Anesthesia will be inducted as before in addition of giving a peribulbar block up to 5 ml (according to the volume of the eye) of Mepivacaine 3% mixed with 10IU of Hyaluronidase by a single injection technique.
  Interventions: Drug: mepivacaine

INTERVENTIONS:
Drug: Articaine and Epinephrine Only Product — comparison between its effect with the other two local anesthetic drugs in peribulbar block on oculocardiac reflex intraoperatively and postoperative pain in pediatrics undergoing squint surgeries with general anesthesia
  Arms: For group A
Drug: levobupivacaine — comparison between its effect with the other two local anesthetic drugs in peribulbar block on oculocardiac reflex intraoperatively and postoperative pain in pediatrics undergoing squint surgeries with general anesthesia
  Arms: Group L
Drug: mepivacaine — comparison between its effect with the other two local anesthetic drugs in peribulbar block on oculocardiac reflex intraoperatively and in peribulbar block on postoperative pain in pediatrics undergoing squint surgeries with general anesthesia
  Arms: Group M

SUMMARY:
To compare the effect of the used local anesthetics in this study on decreasing the incidence of oculocardiac reflex . To evaluate the efficacy of Articaine 4 % , mepivacaine 3% and lidocaine 2% regarding post- operative analgesia.

DETAILED DESCRIPTION:
Population of study: Children undergoing strabismus surgery aged from 7 to 14 years .

* 55 participants grouped randomly into 3 groups :
* Group A :will receive General Anesthesia combined with Peribulbar Block with 5ml of Articaine 4% with 1/100000 adrenaline and 10 International Units (IU) of Hyaluronidase .
* Group L :will receive General Anesthesia combined with Peribulbar Block with 5ml of Lidocaine 2% and 10 IU of Hyaluronidase .
* Group M : will receive General Anesthesia combined with Peribulbar Block with 5 ml of mepivacaine 3% and 10 IU of Hyaluronidase
* Methodology in details:

After obtaining informed written consent from the parents of children after explaining the procedure to them, random allocation of patients into three groups will be done.

In all groups: upon arrival to the operating room, preoperative sedatives in the form of midazolam 0.05 mg/kg by Intravenous route will be used ,standard monitor including; electrocardiogram (ECG), non-invasive blood pressure and pulse oximeter were attached to the patients. The induction of anesthesia will be by intravenous route .

Insertion of 24-22 Gauge Intravenous (IV) catheter and appropriate size laryngeal mask airway (LMA) will be inserted . Anesthesia will be maintained using 100% oxygen and sevoflurane with spontaneous respiration and capnogram will be attached to obtain continuous measurement of end-tidal carbon dioxide (ETCO2).

For group A : General Anesthesia will be inducted as before in addition of giving a peribulbar block up to 5 ml ( according to the volume of the eye ) of Articaine 4 % with adrenaline 1/100000 mixed with 10IU of Hyaluronidase by a single injection technique: a 26/27 gauge needle will be inserted as far laterally as possible in the inferotemporal quadrant. Once the needle is under the globe, it will be directed along the orbital floor, passing the globe equator to a depth controlled by observing the needle/hub junction reaching the plane of the iris. After negative aspiration for blood, with the globe in primary gaze, and start injection and the injected volume will be guided by digital intraocular pressure. For Group L : General Anesthesia will be inducted as before in addition of giving a peribulbar block up to 5 ml ( according to the volume of the eye ) of Lidocaine 2%mixed with 10IU of Hyaluronidase by a single injection technique. For group M: General Anesthesia will be inducted as before in addition of giving a peribulbar block up to 5 ml (according to the volume of the eye) of Mepivacaine 3% mixed with 10IU of Hyaluronidase by a single injection technique. In all of the three groups Intraoperative continuous monitoring with electrocardiography monitor, pulse oximeter and Capnography will be done, and adequate hydration will be taken care of with IV fluid ringer lactate until the oral intake is allowed. In all Groups :monitoring for the incidence of Oculocardiac reflex will be done within (2-3) mins after induction of general anesthesia and giving the Peribulbar Block which is the time of required for draping and sterilization of the eye, there will be intraoperative monitoring for the incidence of Oculocardiac reflex during eye manipulations , good attention for the depth of anesthesia, any rise or drop in the Heart Rate or the Blood Pressure . Intraoperative analgesics using Fentanyl in a dose of 1 mcg/kg will be given intravenously to the patients.

Prophylaxis against post-operative vomiting will be done using Granisterone in a dose of 0.01 mg/kg by intravenous route . Intraoperative mean arterial blood pressure and heart rate will be recorded immediately after induction , at incision time and every 5 mins till the end of the procedure .

Any incidence of oculocardiac reflex will be recorded regarding its onset and time of occurrence and the associated or causing manipulations along with recording of the way the reflex had been dealt with and any given medications or additional blocks required to interfere with the oculocardiac reflex. Any change in the heart rate more than 20 % than the baseline heart rate will be treated by asking the surgeon to stop and if that interference wasn't efficient, an intravenous dose of Atropine of 0.01 mg/kg will be given to the patients and also the dosing of given Atropine will be recorded. After end of the surgery and discontinuation of anesthesia, patients will be transferred to PACU and observed for about 2 hours in the PACU before discharging them to their wards, immediately after discharge and then every 15 mins with total post-operative evaluation time of 6 hours.

Post-operative recovery will be evaluated by using Aldrete score. The post-operative pain will be assessed by using the VAS scale and it will be assessed every 15 mins and any post-operative pain will be recorded , paracetamol will be given regularly in a dose of 15 mg/ kg every 6-8 hours any additional analgesia will be given to the patient if the vas scale > 3 e.g. NSAIDS will be recorded .

Cases with persistent post-operative emesis will be dealt with by appropriate anti-emetic drugs and recorded. Any complications regarding the Peribulbar block (Hemorrhage, Hematoma, etc.) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA I , II.
* Age from 7 to 14 years old.
* Patients undergoing Strabismus Surgery

Exclusion Criteria:

* Patients with ASA III ,IV.
* Patients with Endophthalmitis , orbital fractures.
* Any Congenital or Cardiac anomalies.
* Patients with history of allergy to local anesthetics.
* Revision Surgeries.
* Refusal of the Surgeon. Refusal of the patients' parents

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
The incidence of Intraoperative oculocardiac reflex. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Salem, MD, Principal Investigator — Research Institute of Ophthalmology
Locations (1):
- Research Institute of Ophthalmology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No